CLINICAL TRIAL: NCT00788840
Title: A 24-week, National, Single-centre, Open-labelled, Randomised, Parallel-group Trial Comparing Energy Expenditure With Insulin Detemir Versus NPH Insulin Using a Basal-bolus Regimen With Insulin Aspart as the Mealtime Insulin in Subjects With Type 2 Diabetes
Brief Title: Detemir Energy Expenditure Study
Acronym: DEES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC/2008/14/FHMS
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Isophane Insulin, Human; Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. Insulatard (Active Comparator)
  Interventions: Drug: Insulatard
- 2. Detemir (Active Comparator)
  Interventions: Drug: Detemir

INTERVENTIONS:
Drug: Insulatard — Insulatard insulin used as long-acting insulin for 16-week treatment phase of study.
  Arms: 1. Insulatard
Drug: Detemir — Detemir insulin used as long-acting insulin in treatment phase of study.
  Other Names: Levemir
  Arms: 2. Detemir

SUMMARY:
This is a study designed to compare the effects of 2 long-acting insulins, detemir and insulatard, on energy expenditure,weight, fat composition, gut hormone profiles, glycaemic control and fat and muscle gene expression over a 6 month period.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes
2. Treated with metformin
3. Already on treatment with a long-acting or intermediate insulin.
4. Over 18 years of age,
5. HbA1c > 7.0%
6. BMI 27-40
7. Able and willing to perform self-blood glucose monitoring.
8. Able and willing to maintain consistent eating habits throughout the entire trial period.
9. Able and willing to maintain consistent physical activity level during the entire trial period

Exclusion Criteria:

1. Patients on sulphonylureas or thiazolidinediones
2. Proliferative retinopathy that has required acute treatment within the last six months.
3. Impaired hepatic or renal functions.
4. Cardiac problems.
5. Uncontrolled hypertension (treated or untreated).
6. Mental incapacity, unwillingness or a language barrier precluding adequate understanding or co-operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Weight change | 6 months

SECONDARY OUTCOMES:
Energy Expenditure | 6 months
Fat composition | 6 months
Fat & muscle gene expression | 6 months
Glycaemic control | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Russell-Jones, MB BS, Principal Investigator — University of Surrey
Locations (1):
- Cedar Centre, Royal Surrey County Hospital, Guildford, Surrey, United Kingdom

REFERENCES:
- [Derived] Semlitsch T, Engler J, Siebenhofer A, Jeitler K, Berghold A, Horvath K. (Ultra-)long-acting insulin analogues versus NPH insulin (human isophane insulin) for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 9;11(11):CD005613. doi: 10.1002/14651858.CD005613.pub4. PMID 33166419